CLINICAL TRIAL: NCT06563336
Title: Effects of the EMG-driven Hand Robot Training in Patients With Hand Dysfunction Due to Nerve Damage From Burns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HangangSHH-19
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Burn Hand; Rehabilitation
Keywords: hand burn; robot training; hand functions; skin characteristics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measurements were performed at baseline and immediately after 12 weeks rehabilitation. The outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG-driven hand robot training (Experimental): Robot rehabilitation program was applied with Hand of Hope®(Rehab-Robotics Company, Hong Kong), and EMG-driven exoskeleton. The biggest advantage of this system is that it measures the residual muscle activity values with surface EMG(sEMG) sensors. The residual muscles activity is used by giving feedback to the patient.
  Participants in the experimental group and the control group received 60 sessions of hand rehabilitation programs delivered 5 times a week over 12 weeks. Experimental group performed robotic rehabilitation for 30 minutes and conventional occupational treatment for 30 minutes a day.
  Interventions: Other: EMG-driven hand robot training; Other: conventional occupational training
- conventioanl training (Active Comparator): The control group performed 30-minutes conventional occupational treatment twice a day. In both groups, the hand rehabilitation program was carried out at the same time and interval for 60 minutes a day.
  Interventions: Other: conventional occupational training

INTERVENTIONS:
Other: EMG-driven hand robot training — Robot rehabilitation program was applied with Hand of Hope®(Rehab-Robotics Company, Hong Kong), and EMG-driven exoskeleton. The biggest advantage of this system is that it measures the residual muscle activity values with surface EMG(sEMG) sensors. The residual muscles activity is used by giving feedback to the patient.
  This treatment program, which was applied to both groups in the study, consisted of joint range of motion (ROM) exercises, stretching exercises for burn scars, strengthening exercises using putty or bands, and fine motor training such as writing and using a chopstick.
  Arms: EMG-driven hand robot training
Other: conventional occupational training — This treatment program, which was applied to both groups in the study, consisted of joint range of motion (ROM) exercises, stretching exercises for burn scars, strengthening exercises using putty or bands, and fine motor training such as writing and using a chopstick.

SUMMARY:
Hands are the most frequent burn injury sites. Appropriate rehabilitation is essential to ensure good functional recovery. The aim of this study was to investigate the effects of EMG driven robotic rehabilitation on hand functions and skin characteristics of patients with nerve damage caused by burns. A randomized controlled, single blind trial recruited the patients with hand dysfunction after burn injury. The participants were randomly allocated to experimental group (EG) and control group (CG) for 5 days a week and totally 60 sessions for 12 weeks. The EG received robotic assisted hand training with the EMG-driven exoskeleton hand robot (Hand of Hope®.Rehab-Robotics Company) and conventional occupational therapy. The CG performed conventional occupational therapy, including hand range of motion (ROM) exercises and hand functional training twice a day for 12 weeks. Outcome measures were as follows: 10-point visual analog scale for pain, Jebsen-Taylor hand function test, grip strength, Purdue Pegboard test, joint ROMs, ultrasound measurement of scar thickness, and skin characteristics before and immediately after 12 weeks of treatment. There is still no established protocol for burn injury rehabilitation. The aim of this study was to investigate the effects of EMG driven robotic rehabilitation on hand functions and skin characteristics of patients with nerve damage and scarring caused by burns.

DETAILED DESCRIPTION:
The hand represents the area of the body most common affected by burns, accounting for 80% of all burn injuries. The deformities and scarring that occur when the affected area is the hand can result in the loss of function such as grip strength, range of motion (ROM), dexterity. While early excision and grafting have been shown to reduce the loss of function in cases of burns, up to 30% of affected joints have been found to have a limited ROM.Acute hand rehabilitation tailored to the patient's condition is essential after a burn injury.However, there is still no proven hand rehabilitation protocol in burn centers, new rehabilitation modalities are being attempted to improve hand function.Robot training is being attempted to improve function in musculoskeletal diseases including burns,and the researchers have confirmed the clinical effectiveness of applying a soft glove-type hand robot for hand burns.There is still no established protocol for burn injury rehabilitation. This study was designed as a prospective, randomized controlled single-blind, case control study. The participants were randomly allocated to experimental group (EG) and control group (CG) for 5 days a week and totally 60 sessions for 12 weeks. The EG received robotic assisted hand training with the EMG-driven exoskeleton hand robot (Hand of Hope®.Rehab-Robotics Company) and conventional occupational therapy. The CG performed conventional occupational therapy, including hand range of motion (ROM) exercises and hand functional training twice a day for 12 weeks. Outcome measures were as follows: 10-point visual analog scale for pain, Jebsen-Taylor hand function test, grip strength, Purdue Pegboard test, joint ROMs, ultrasound measurement of scar thickness, and skin characteristics before and immediately after 12 weeks of treatment. The aim of this study was to investigate the effects of EMG driven robotic rehabilitation on hand functions and skin characteristics of patients with nerve damage and scarring caused by burns.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* more than 50% of the hand is burned
* burns occurred on the right hand, which is the dominant hand
* had a deep partial-thickness (second-degree) or a full-thickness (third-degree) burn, which had been treated with a split-thickness skin graft (STSG) after the burn injury
* nerve injury to the hand was confirmed by electromyography
* all patients were in the re-epithelialization phase

Exclusion Criteria:

* other causes of musculoskeletal diseases (rheumatoid arthritis and degenerative joint diseases et al) that may affect hand dysfunctions
* unstable scars (acute infection or coagulopathy) that may cause damage to the scar area during hand treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
A 10-point visual analog scale (VAS) | 12 weeks
  was used to measure the scar pain severity, with ratings ranging from 0 (no pain) to 10 (unbearable pain).

SECONDARY OUTCOMES:
Patients were assessed using the total active motion (TAM) | 12 weeks
  The sum of the angles of flexion and extension of the metacarpophalangeal joint, proximal interphalangeal joint, and distal interphalangeal joint of each finger. A maximum of 260 degrees to a minimum of -260 degrees for each finger.
Jebsen-Taylor hand function test (JTT) | 12 weeks
  performance speed of standardized seven tasks, each scored on a 0-15-point scale (with higher scores indicating better hand function)
the Purdue Pegboard test (PPT) | 12 weeks
  motor function was measured as the number of pins that could be placed on the board in 30 s, with dextrity measured as the number of pins, washers, and collars that could be assembled in 60 s
Scar thickness | 12 weeks
  was objectively quantified using ultrasonography (128 BW1 US system, Medison, Korea).
Trans-epidermal water loss (TEWL) | 12 weeks
  was measured using a Tewameter® (Courage-Khazaka Electronic GmbH, Germany) to evaluate water evaporation.Higher numbers mean drier skin.
erythema and pigmentation | 12 weeks
  Mexameter®(MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure the melanin levels and the severity of erythema. Higher values mean more pigmentation and reddness.
Sebum | 12 weeks
  was measured with the Sebumeter® (Courage-Khazaka Electronic GmbH, Germany). The microprocessor calculated the results, which were on display, in mg/cm2.
Distensibility | 12 weeks
  measured using Cutometer SEM 580® (Courage-Khazaka Electronic GmbH, Cologne, Germany). Two seconds of negative pressure at 450 mbar was followed by 2 s of recess, which consisted of a complete cycle.The higher the measurement value, the better the expansion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang sacred heart hodpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Padilla-Castaneda MA, Sotgiu E, Barsotti M, Frisoli A, Orsini P, Martiradonna A, Laddaga C, Bergamasco M. An Orthopaedic Robotic-Assisted Rehabilitation Method of the Forearm in Virtual Reality Physiotherapy. J Healthc Eng. 2018 Aug 1;2018:7438609. doi: 10.1155/2018/7438609. eCollection 2018. PMID 30154992
- [Result] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552